CLINICAL TRIAL: NCT00469417
Title: A Multicenter, Phase III, Randomised Study of Photodynamic Therapy With Metvix Cream 160 mg/g in Comparison With Cryotherapy in Patients With Primary Superficial Basal Cell Carcinoma
Brief Title: Metvix Photodynamic Therapy (PDT) Versus Cryotherapy in Participants With Primary Superficial Basal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC T304/99
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Superficial Basal Cell Carcinoma
Keywords: Methyl aminolevulinate; Photodynamic therapy; Primary Superficial Basal Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metvix® PDT (Experimental): Participants with basal cell carcinoma (BCC) lesions were administered to photodynamic therapy (PDT) with Metvix® cream 160 milligrams per gram (mg/g) applied for three hours, followed by illumination using non-coherent light with a fluency of 75 Joule per centimeter square (J/cm*2) and fluency rate of 70-200 milliwatt per centimeter square (mW/cm*2) up to 13 weeks.
  Interventions: Drug: Metvix® cream
- Cryotherapy (Active Comparator): Cryotherapy was performed with a hand-held liquid nitrogen spray, using a double freeze-thaw cycle. After an initial icefield formation with a 3 millimeter (mm) rim of clinically healthy tissue, the icefield was to be maintained for a minimum of 20 seconds. This procedure was repeated after a thaw of 2-3 times the freeze time up to 12 weeks.
  Interventions: Procedure: Hand held liquid nitrogen spray cryotherapy

INTERVENTIONS:
Drug: Metvix® cream
  Other Names: Methyl 5-aminolevulinate hydrochloride
  Arms: Metvix® PDT
Procedure: Hand held liquid nitrogen spray cryotherapy
  Arms: Cryotherapy

SUMMARY:
The purpose of this study was to compare the efficacy of Photodynamic Therapy (PDT) methyl aminolevulinate (MAL) cream to cryotherapy, in treatment of participants with primary superficial basal cell carcinoma (BCC).

Secondary objectives was to compare cosmetic outcome and tolerability (adverse events) in these participants, 3 months after treatment. In addition the recurrence rates in the two treatment groups will be compared up to five years after treatment.

DETAILED DESCRIPTION:
BCC was a highly frequent skin malignancy, and accounts for approximately 75% of all non-melanoma skin cancers. It is the most common malignant tumour of any organ, mostly affecting head and neck (84%) in fair-skinned people. Several non-pharmacological treatment modalities was used for BCC, including excision surgery, Moh's surgery, radiation, curettage/electrodesiccation and cryotherapy. The treatment used depends on the type, size, depth and localisation of the BCC lesion.

The use of PDT was attractive for the treatment of BCCs because of its efficiency, mild and local side effects and excellent cosmetic outcome. Previous clinical experience was promising and participants with primary BCCs were included in this prospective, randomised, comparative, multicenter study to show that Metvix is non-inferior to alternative treatment with better cosmetic outcome.

The primary end-point is the number of participants in whom 75% or more of the BCC lesions have responded completely at 3 months after PDT with Metvix or 3 months after cryotherapy. Both on-site and independent, blinded response assessments analysed. The analysis based on the results of the independent review board constitutes the primary analysis.

The secondary end-points was the proportion of participants in whom less than 75% of the BCC lesions respond completely, number of lesions across participants that show complete response, evaluation of cosmetic outcome and adverse events 3 months after Metvix PDT or 3 months after cryotherapy. In addition 12, 24, 36, 48 and 60 months recurrence rates was assessed.

ELIGIBILITY:
Inclusion Criteria:

A participant with superficial BCC lesion(s) suitable for entry was defined as a participant with:

* histologically confirmed diagnosis of primary superficial BCC lesion(s)
* BCC lesions suitable for cryotherapy
* males or females above 18 years of age
* written informed consent. In accordance with Amendment 2 (local amendment), only participant above 19 years of age were to be included in Austria.

Exclusion Criteria:

A participant or lesion fulfilling any of the following criteria was ineligible for inclusion:

* prior treatment of the BCC lesion(s)
* participant with more than 10 eligible BCC lesions
* a superficial BCC lesion with the largest diameter exceeding 15 mm on face/scalp, larger than 20 mm on extremities and neck and larger than 30 mm on the trunk
* a superficial BCC lesion with the largest diameter smaller than 6 mm
* participant with porphyria
* participant with Gorlin's syndrome
* pigmented superficial BCC lesion(s)
* morpheaform lesion(s)
* infiltrating lesion(s)
* participants with a history of arsenic exposure
* known allergy to Metvix®, a similar PDT compound or excipients of the cream
* participation in other clinical studies either concurrently or within the last 30 days
* pregnant or breast-feeding; all women of child-bearing potential had to document a negative pregnancy test and use the pill or intrauterine device during the treatments and for at least one month thereafter
* conditions associated with a risk of poor protocol compliance.

In Amendment 1 the following exclusion criteria were added:

* xeroderma pigmentosum lesion
* concurrent use of immunosuppressive medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1999-10-18 (Actual); Primary Completion 2001-09-05 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Basset-Séguin, Professor, Principal Investigator — Saint-Louis Hospital, Paris
Locations (14):
- University of Graz, Graz, Austria
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Helsinki University Central Hospital, Helsinki, Finland
- France (2):
  - Hôpital Sainte-Marguerite, Marseille
  - Service de Dermatologie, C.H.U Saint Louis, Paris
- Spedali di Brescia, Brescia, Italy
- Sweden (4):
  - Länsjukhuset Ryhov, Jönköping
  - Universitetssjukhuset, Linköping
  - Regionsjukhuset i Örebro, Örebro
  - Huddinge Sjukhus, Stockholm
- United Kingdom (4):
  - University of Wales, Cardiff
  - Ninewells Hospital, Dundee
  - Falkirk and District Royal Infirmary, Falkirk
  - Glasgow University Hospital, Glasgow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 120 participants were randomized, of which 118 were received the study treatment. The study was carried out in 13 centers in seven European countries, they were included (Sweden, Finland, United Kingdom, Austria, France, Belgium and Italy).
Period: Overall Study
Arm/Group | Metvix® PDT | Cryotherapy
Started | 62 | 58
Treated | 60 | 58
Completed | 32 | 41
Not Completed | 30 | 17
Not completed — Treatment failure all lesions | 18 | 11
Not completed — Consent withdrawn | 1 | 1
Not completed — Adverse Event | 8 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Intercurrent disease | 0 | 1
Not completed — Randomized but not treated | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis set included all the participants enrolled in the study who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metvix® PDT | Cryotherapy | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (16) | 64 (13) | 64 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 40 | 30 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 60 | 58 | 118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Histologically Confirmed Patient Complete Response (CR) 3 Months After Last Metvix PDT or Cryotherapy Cycle
Description: Patient Complete Response (CR) was defined as 100 percentage of the lesions within the participant having negative findings for nodular basal cell carcinoma (BCC) in the histological examination.
Time Frame: 3 months after last Metvix PDT or Cryotherapy cycle, up to 6 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Metvix® PDT | Cryotherapy
Number analyzed (Participants) | 60 | 58
percentage of participants | 92 | 90

2. Secondary Outcome: Number of Lesion With Complete Response 3 Months After Last Metvix PDT or Cryotherapy Cycle
Description: Complete response was defined as no clinically visible BCC lesions in the treatment area.
Time Frame: 3 months after last Metvix PDT or Cryotherapy cycle, up to 6 months
Population: as for baseline characteristics
Measure: Number; unit: lesion
Units Other Than Participants: lesion
Arm/Group | Metvix® PDT | Cryotherapy
Number analyzed (Participants) | 60 | 58
Number analyzed (lesion) | 114 | 105
lesion | 109 | 94

3. Secondary Outcome: Overall Cosmetic Outcome Assessed by Investigator 3 Months After the Last Metvix PDT or Cryotherapy Cycle
Description: Cosmetic outcome was assessed by both investigator and participants in participants with 100% of lesions in complete response. Overall cosmetic outcome was assessed with regard to occurrence of the following signs or symptoms; scarring, atrophy, induration, redness or change in pigmentation. The investigator graded the cosmetic outcome as:
  * excellent: no scarring, atrophy or induration, and no or slight occurrence of redness or change in pigmentation compared lo adjacent skin
  * good: no scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin
  * fair: slight to moderate occurrence of scarring, atrophy or induration
  * poor: extensive occurrence of scarring, atrophy or induration.
Time Frame: 3 months after the last metvix PDT or Cryotherapy cycle (Up to 6 months)
Population: Intent-to-treat analysis set included all the participants enrolled in the study who received at least one dose of study treatment. Here overall "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix® PDT | Cryotherapy
Number analyzed (Participants) | 53 | 50
Participants
  Investigator: Excellent | 17 | 2
  Investigator: Good | 30 | 23
  Investigator: Fair | 6 | 25

4. Secondary Outcome: Overall Cosmetic Outcome Assessed by Participants 3 Months After the Last Metvix PDT or Cryotherapy Cycle
Description: Cosmetic outcome was assessed by both investigator and participants in participants with 100% of lesions in complete response. Overall cosmetic outcome was assessed with regard to occurrence of the following signs or symptoms; scarring, atrophy, induration, redness or change in pigmentation. The participants graded the cosmetic outcome as:
  * excellent: no scarring, atrophy or induration, and no or slight occurrence of redness or change in pigmentation compared lo adjacent skin
  * good: no scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin
  * fair: slight to moderate occurrence of scarring, atrophy or induration
  * poor: extensive occurrence of scarring, atrophy or induration.
Time Frame: 3 months after the last metvix PDT or Cryotherapy cycle (Up to 6 months)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix® PDT | Cryotherapy
Number analyzed (Participants) | 46 | 44
Participants
  Participants: Excellent | 22 | 9
  Participants: Good | 24 | 24
  Participants: Fair | 0 | 11

5. Secondary Outcome: Recurrence Rate in Complete Clearance Group
Description: Recurrence rate in complete clearance group was analyzed.
Time Frame: 12, 24, 36, 48 and 60 months after last Metvix PDT cycle or Cryotherapy (Up to 5 years)
Population: Intent-to-treat analysis set included all the participants enrolled in the study who received at least one dose of study treatment. Here "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: lesion
Units Other Than Participants: lesion
Arm/Group | Metvix® PDT | Cryotherapy
Number analyzed (Participants) | 55 | 52
Number analyzed (lesion) | 109 | 94
lesion
  12 months | 10 | 12
  24 months | 18 | 18
  36 months | 23 | 18
  48 months | 23 | 18
  60 months | 23 | 19

6. Secondary Outcome: Overall Cosmetic Outcome Assessed by Investigator 24, 36, 48, and 60 Months After the Last Metvix PDT or Cryotherapy Cycle
Description: as for outcome 3
Time Frame: 24, 36, 48, and 60 Months After the Last Metvix PDT Cycle (Up to 5 years)
Population: Intent-to-treat analysis set included all the participants enrolled in the study who received at least one dose of study treatment. Here overall "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure. "Number analyzed", signifies those participants who were evaluable for this outcome measure at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix® PDT | Cryotherapy
Number analyzed (Participants) | 36 | 43
Participants
  Excellent: At month 24: number analyzed (Participants) | 34 | 38
  Excellent: At month 24 | 19 | 3
  Good: At month 24: number analyzed (Participants) | 34 | 38
  Good: At month 24 | 12 | 15
  Fair: At month 24: number analyzed (Participants) | 34 | 38
  Fair: At month 24 | 3 | 20
  Excellent: At month 36 | 20 | 5
  Good: At month 36 | 12 | 22
  Fair: At month 36 | 4 | 14
  Poor: At month 36 | 0 | 2
  Excellent: At month 48: number analyzed (Participants) | 33 | 42
  Excellent: At month 48 | 19 | 5
  Good: At month 48: number analyzed (Participants) | 33 | 42
  Good: At month 48 | 10 | 21
  Fair: At month 48: number analyzed (Participants) | 33 | 42
  Fair: At month 48 | 4 | 15
  Poor: At month 48: number analyzed (Participants) | 33 | 42
  Poor: At month 48 | 0 | 1
  Excellent: At month 60: number analyzed (Participants) | 32 | 43
  Excellent: At month 60 | 18 | 6
  Good: At month 60: number analyzed (Participants) | 32 | 43
  Good: At month 60 | 8 | 22
  Fair: At month 60: number analyzed (Participants) | 32 | 43
  Fair: At month 60 | 6 | 14
  Poor: At month 60: number analyzed (Participants) | 32 | 43
  Poor: At month 60 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Months 60
Description: Safety analysis set included all the participants enrolled in the study.
Arm/Group | Metvix® PDT | Cryotherapy
All-Cause Mortality (participants affected / at risk) | 4/60 | 3/58
Serious Adverse Events (participants affected / at risk) | 7/60 | 2/58
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metvix® PDT (N=60) | Cryotherapy (N=58)
Death due to myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Metastatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Participant deceased (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic adenocarcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes